CLINICAL TRIAL: NCT02708355
Title: A Pilot Phase IV, Multicenter, Randomized, Double Blind, Placebo-Controlled, Parallel Study To Investigate The Correlation Between Ph Control And Heartburn Symptoms After 14 Days Of Proton Pump Inhibitor Treatment In Subjects With Frequent Heartburn
Brief Title: Pilot Study To Investigate The Association Between Acid Control And Heartburn Symptoms After Proton Pump Inhibitor Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: B5141005; ACID CONTROL EXPLORATORY STUDY (Other: Alias Study Number)
Record Dates: First submitted 2016-01-21; First posted 2016-03-15 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Heartburn
MeSH Terms: conditions — Heartburn | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Esomeprazole 20 mg once daily (Experimental): Esomeprazole 20 mg administered orally in the morning and placebo administered orally in the evening
  Interventions: Drug: Esomeprazole 20 mg; Drug: Placebo
- Esomeprazole 20 mg twice daily (Experimental): Esomeprazole 20 mg administered orally in the morning and esomeprazole 20 mg administered orally in the evening
  Interventions: Drug: Esomeprazole 20 mg
- Placebo (Placebo Comparator): Placebo administered orally in the morning and placebo administered orally in the evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole 20 mg — Esomeprazole 20 mg banded capsules (22.3 mg esomeprazole magnesium trihydrate)
  Other Names: Nexium
  Arms: Esomeprazole 20 mg once daily; Esomeprazole 20 mg twice daily
Drug: Placebo — Placebo capsules
  Arms: Esomeprazole 20 mg once daily; Placebo

SUMMARY:
The purpose of this pilot study is to investigate the association between gastric acid suppression and relief of 24 hour heartburn following treatment with the proton pump inhibitor (PPI) drug esomeprazole in frequent heartburn patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed symptom history of heartburn, acid regurgitation, or epigastric pain of at least 3 months, while treating with gastric acid modulating therapy (antacids, H2 receptor antagonists (H2RAs) and/or PPIs).
* Heartburn symptoms that average 3 times per week or greater including at least 2 episodes of nighttime heartburn symptoms per week over the past 30 days.
* When heartburn medications were used, subject had heartburn symptoms that were responsive to antacids, non prescription H2RAs, or short term non prescription or prescription PPIs at approved doses but complete resolution of heartburn was not achieved.

Exclusion Criteria:

* A history (past or present) of erosive esophagitis verified by endoscopy.
* The need for continuous treatment with H2RAs, PPIs, gastric prokinetic drugs, or antacids for any indication through the study (eg, long term prescription therapy).
* Subjects requiring continuous intervention by a physician for the treatment of GERD (ie, treatment of erosive esophagitis or prevention of relapse of healed esophagitis).

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - St. Anthony Hospital - Conference Rooms, Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Miner PB, Johnson DA, Katz PO, Li J, Gatoulis SC, Pollack C. Pilot, Randomized, Blinded, Placebo-Controlled Trial Investigating the Correlation Between Acid Control and Heartburn Relief with 14 Days of Esomeprazole Treatment. Adv Ther. 2018 Nov;35(11):2024-2040. doi: 10.1007/s12325-018-0792-z. Epub 2018 Sep 25. PMID 30255418
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5141005&StudyName=A%20Pilot%20Phase%20Iv%2C%20Multicenter%2C%20Randomized%2C%20Double%20Blind%2C%20Placebo-controlled%2C%20Parallel%20Study%20To%20Investigate%20The%20Correlation%20Between%20Ph%20Control%20And%20Heartburn%20Symptoms%20After%2014%20Days%20Of%20Proton%20Pump%20Inhibitor%20Treatment%20In%20Subjects%20With%20Frequent%20Heartburn
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5141005&StudyName=A+Pilot+Phase+Iv%2C+Multicenter%2C+Randomized%2C+Double+Blind%2C+Placebo-controlled%2C+Parallel+Study+To+Investigate+The+Correlation+Between+Ph+Control+And+Heartburn+Symptoms+After+14+Days+Of+Proton+Pump+Inhibitor+Treatment+In+Subjects+With+Frequent+Heartburn

RESULTS

PARTICIPANT FLOW:
Groups:
- Esomeprazole 20 mg Twice Daily: Esomeprazole 20 milligram capsules administered orally twice daily from Day 1 to 14.
- Esomeprazole 20 mg Once Daily + Placebo: Esomeprazole 20 mg capsule administered orally once daily in the morning and placebo matched to esomeprazole capsule once daily in the evening from Day 1 to 14.
- Placebo: Placebo matched to esomeprazole capsules administered orally twice daily from Day 1 to 14.
Period: Overall Study
Arm/Group | Esomeprazole 20 mg Twice Daily | Esomeprazole 20 mg Once Daily + Placebo | Placebo
Started | 21 | 22 | 12
Completed | 20 | 22 | 12
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole 20 mg Twice Daily | Esomeprazole 20 mg Once Daily + Placebo | Placebo | Total
Number analyzed (Participants) | 21 | 22 | 12 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (10.23) | 40.8 (10.95) | 44.7 (10.50) | 41.9 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 9 | 34
  Male | 10 | 8 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relief of 24 Hour Heartburn and Without Relief of 24 Hour Heartburn
Description: Relief of 24 hour heartburn was defined as a daily diary response of "0" to the question "Over the last 24 hours (yesterday and last night), what was the severity of your most intense episode of heartburn?" on at least 6 of the participant's last 7 consecutive days [Days 8 - 14] of treatment allowing for one day with a maximum severity of "2".The response was noted by participants in the diary for last 7 consecutive days [Day 8 - 14] on a 3 point scale ranged from 0 to 2 where 0= complete relief and 2= maximum severity. Higher score indicated worse condition/more severity. In this outcome measure, participants with relief of 24 hour heartburn and participants without relief of 24 hour heartburn were reported.
Time Frame: Day 8 up to Day 14
Population: Per protocol analysis set included all randomized participants who provided valid data for Day -1 PH monitoring, take at least one dose of randomized study medication, complete the 14 day treatment phase, undergo and provide valid data for Day 14 pH monitoring and complete at least 5 days of diary entries in each of Days -7 to -1 and Days 8 to 14.
Measure: Number; unit: participants
Arm/Group | Esomeprazole 20 mg Twice Daily | Esomeprazole 20 mg Once Daily + Placebo | Placebo
Number analyzed (Participants) | 16 | 18 | 5
participants
  With Relief | 7 | 10 | 0
  Without Relief | 9 | 8 | 5

2. Primary Outcome: Change From Baseline at Day 14 in Percentage of Time Over 24--Hour Period With Intra Gastric pH Greater Than (>)4
Description: Percentage of time was calculated over the 24 hour period during which intra gastric pH >4 was observed. Relief of 24 hour heartburn was defined as a daily diary response of "0" to the question "Over the last 24 hours (yesterday and last night), what was the severity of your most intense episode of heartburn?" on at least 6 of the participant's last 7 consecutive days [Days 8 - 14] of treatment allowing for one day with a maximum severity of "2".The response was noted by participants in the diary for last 7 consecutive days [Day 8 - 14] on a 3 point scale ranged from 0 to 2 where 0= complete relief and 2= maximum severity. Higher score indicated worse condition/more severity. In this outcome, change from baseline at Day 14 in percentage of time over the 24 hour period during which intra gastric pH >4 was observed, was reported.
Time Frame: Baseline, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Esomeprazole 20 mg Twice Daily | Esomeprazole 20 mg Once Daily + Placebo | Placebo
Number analyzed (Participants) | 16 | 18 | 5
percentage of time
  Baseline | 12.53 (18.045) | 13.35 (9.069) | 12.32 (5.635)
  Change at Day 14 | 70.23 (23.105) | 42.83 (18.654) | 0.78 (5.839)
Statistical Analysis 1: Comparison: Esomeprazole 20 mg Twice Daily vs Esomeprazole 20 mg Once Daily + Placebo vs Placebo; Association between percentage of time with intragastric pH>4 and relief of 24 -hour heartburn was assessed using logistic regression model with relief of 24- hour heartburn at Day 14 as dependent variable and change in percentage of time with intragastric pH>4 as the independent variable, controlling for age, sex, and body mass index (BMI); Test type: Superiority or Other; p = 0.0442, Regression, Logistic; Odds Ratio (OR) = 1.028, 95% CI 2-sided [1.001 to 1.055]

ADVERSE EVENTS:
Arm/Group | Esomeprazole 20 mg Twice Daily | Esomeprazole 20 mg Once Daily + Placebo | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/12
Other Adverse Events (participants affected / at risk) | 3/21 | 1/22 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 20 mg Twice Daily (N=21) | Esomeprazole 20 mg Once Daily + Placebo (N=22) | Placebo (N=12)
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.